CLINICAL TRIAL: NCT03498755
Title: The Invisible Fishers: Empowering and Safeguarding Women in Fisheries Value Chains in Ghana to Reduce Anemia
Brief Title: The Invisible Fishers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Ghana (Other); Innovations for Poverty Action (Other); Netherlands Development Organization (Unknown); Viamo (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Andrew Jones, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00138934
Record Dates: First submitted 2018-03-12; First posted 2018-04-17 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Anemia
Keywords: fisheries; Ghana; sub-Saharan Africa; value chain; fish processing; fish smoking
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Two communities in each of two study regions will be assigned to one of the three treatments (i.e., six communities in total per region). Assigning two communities to the same treatment in each region will allow us to assess differential intervention design and implementation needs for communities in similar geographic areas. Ten women in each community will be purposefully selected for participation to ensure intra-community variation on participant age, socioeconomic status, years of experience with fish smoking, and the scale of fish smoking enterprises. Across both regions, 120 women will be recruited from a total of 12 communities. While the interventions will be delivered to individual women, treatment assignment will be carried out at the community-level given the risk of sharing information and inputs within communities that could contaminate intervention exposure and bias observed treatment effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multi-sectoral anemia behavior change (Experimental): Address multiple behavioral determinants of anemia by promoting the identification, knowledge, valuation and practice of four behavioral domains: 1) consumption of micronutrient-rich animal-source foods; 2) malaria and soil-transmitted helminth infection control practices; 3) water, sanitation and hygiene (WASH) best practices; and 4) women's autonomy in decision-making and control of the use of earned income.
  Interventions: Behavioral: Mobile phone audio messaging; Behavioral: Peer-to-peer learning
- Strengthening market engagement of fish processors (Experimental): Assist women in overcoming limited access to credit, inadequate storage facilities, and insufficient information about market prices, which constrain the timeliness and amount of market-ready product available for sale, through a three-pronged approach that includes: 1) a conditional cash transfer; 2) entrepreneurship training; and 3) enhanced access to market price information.
  Interventions: Behavioral: Mobile phone audio messaging; Behavioral: Peer-to-peer learning; Behavioral: Conditional cash transfer; Behavioral: Entrepreneurship training; Behavioral: Market price information
- Improving fish smoking technology and practices (Experimental): Introduce and promote a recently developed fish smoking oven known as the Ahotor, which was explicitly designed to reduce emission from biomass fuel combustion, decrease polycyclic aromatic hydrocarbon (PAH) levels of smoked fish, and increase fuel efficiency. Use of this oven will reduce workload, increase earnings, and reduce harmful occupational exposures. Introduction of this improved fish smoking oven will be combined with behavior change education focused on promoting optimal fish smoking and handling practices.
  Interventions: Behavioral: Mobile phone audio messaging; Behavioral: Peer-to-peer learning; Behavioral: Improved smoke ovens

INTERVENTIONS:
Behavioral: Mobile phone audio messaging — Audio messages will be "pushed" to participants' mobile phones twice weekly on a set schedule in discrete modules that include basic information related to each of the four behavioral domains followed by an integration of the information across behaviors through relatable, character-driven narratives that enable message recipients to engage with the content through a real-world context.
Behavioral: Peer-to-peer learning — Women participants in each community will meet twice monthly for peer-to-peer learning sessions to reinforce the content of audio messages. These sessions will further use women's empowerment approaches including critical examination of gender dynamics, and discussions of solutions for equitable decision-making and control of resources within households. These discussions will be facilitated with male household members and grandmothers in separate learning sessions that will be held three times throughout the intervention period.
Behavioral: Conditional cash transfer — Participants will receive a conditional cash transfer to support their fish smoking business. The payment will be conditional on their participation in entrepreneurship trainings and the use of the investment into their fish smoking business.
  Arms: Strengthening market engagement of fish processors
Behavioral: Entrepreneurship training — Entrepreneurship training will focus on commonly lacking business knowledge, with an emphasis on establishing fundamental entrepreneurial skills (i.e., customer care, accounting), sound business management and decision-making, building strong and sustainable business relationships, and encouraging the use of loans for their intended purposes. This training will be introduced during the credit and savings group (CSG) meetings that will occur twice per month.
  Arms: Strengthening market engagement of fish processors
Behavioral: Market price information — Average market prices for fresh and processed fish at community, district, and regional markets will be disseminated via audio message calls (using Viamo's Infoline platform) to the mobile phones of women with the price information in their preferred language. These market prices will be collected twice weekly by Viamo field enumerators and sent to regional coordinators for validation. A second, independent validation will be carried out to ensure that there are no discrepancies.
  Arms: Strengthening market engagement of fish processors
Behavioral: Improved smoke ovens — Local private sector artisans will construct and serve as suppliers of the new ovens. The promotion, uptake and impact of these improved Ahotor ovens will be tested among study participants. Awareness-raising workshops held in each community will promote the Ahotor in concert with a public retrofitting of a Chorkor stove. Immediately following this event, one month later, and three months later, study participants will receive additional one-on-one counseling to provide further support on the proper use of the smoke oven, as well as on optimal handling and smoking practices to enhance product quality.
  Arms: Improving fish smoking technology and practices

SUMMARY:
This pilot study aims to introduce three interventions directed toward mitigating anemia among women in Ghana, including: 1) multi-sectoral behavior change, 2) strengthening market engagement of fish processors, 3) improving fish smoking technology and practices. These interventions will be implemented among female fish processors, a population that represents a promising focal area for intervention within fisheries value chains, which have been identified as a uniquely promising sector for intervention to mitigate anemia among women. The investigators expect that the findings from this study will inform understanding of how best to design, implement, and evaluate interventions into fisheries and other animal-source food value chains in Ghana and across sub-Saharan Africa to address anemia and other nutritional and health concerns.

DETAILED DESCRIPTION:
Anemia among women of reproductive age remains an intractable public health problem in many low- and middle-income countries, especially in sub-Saharan Africa (SSA) where more than one-third of women of reproductive age are anemic. The complex etiology of anemia suggests the importance of designing interventions that address both nutritional deficiencies and environmental drivers of anemia risk. This proposed research builds on new knowledge generated from ongoing formative research by our investigator team aimed at understanding the potential for interventions into animal-source food (ASF) value chains to influence anemia among adolescent girls and women in Ghana. The investigators have identified fisheries value chains in Ghana as a uniquely promising sector for intervention to mitigate anemia among women. Specifically, our research indicates that fish processing is the most promising focal area for intervention within fisheries value chains to address anemia among women. Therefore, the overall research objective of this proposed research is to develop, adapt, and pilot test a set of interventions into fisheries value chains in Ghana aimed at mitigating anemia among women. Specifically, the investigators aim to: 1) define the scope, feasibility, and scalability of priority intervention strategies that have been identified through our ongoing formative research, 2) adapt the interventions to the proposed study contexts, and 3) design and pilot test specific implementation strategies, as well as a monitoring and evaluation (M&E) framework for assessing intervention delivery, uptake, impacts, and mechanisms of impact at multiple loci along hypothesized program impact pathways.

Our ongoing formative research and an extended consultation process with stakeholders and community participants have identified priority strategies for intervention within fisheries value chains in Ghana that are feasible, scalable, likely to reduce anemia through multiple mechanisms, and for which there is clear potential for sustainability of impact. The investigators expect that the pilot testing of these interventions and the associated M&E framework will directly inform the design, implementation and evaluation of a full randomized controlled trial (RCT) that will evaluate the effectiveness of these interventions on anemia mitigation among women in Ghana. As such, the design of this pilot research will mimic that of a RCT with three distinct treatments delivered to women in separate study arms, each arm reflecting the priority intervention strategies identified through our ongoing formative research:

* Treatment Arm 1 (TA1): a multi-sectoral anemia behavior change intervention focused on promoting a diversity of anemia-mitigating behaviors including consumption of micronutrient-rich ASFs, malaria and soil-transmitted helminth control practices, and water, sanitation and hygiene best practices (TA1 is also a component of Treatment Arms 2 and 3);
* Treatment Arm 2 (TA2): an intervention aimed at strengthening women fish processors' engagement with markets through a group-based microcredit scheme, providing entrepreneurship training, and facilitating enhanced access to market price information;
* Treatment Arm 3 (TA3): an intervention introducing improved fish smoking technology and practices to women processors aimed both at improving earnings and reducing harmful occupational exposures associated with fish smoking.

The investigators will recruit a total of 120 total participants from 12 communites in two regions of Ghana that represent marine and fresh water small-scale fisheries systems. Participants will be recruited into a nine-month pilot intervention with data collection occurring at baseline prior to the start of the intervention, at the middle point of intervention implementation, and at endline immediately following completion of intervention implementation. The investigators will use survey-based instruments, direct observation, participant diaries, anthropometric and dietary assessment, occupational exposure assessment, as well as analysis of blood and stool specimens to evaluate changes in anemia, micronutrient status, inflammation and infection, as well as changes in participants' knowledge, attitudes, behaviors, and exposures that the investigators hypothesize are linked to intervention exposure. Such an analysis is critical for understanding the relative importance of different mechanisms of impact for each intervention. The investigators will further carry out qualitative, semi-structured interviews with study participants and project implementation staff to understand their perceptions of the interventions, factors that facilitated or prevented successful implementation and uptake of interventions, and their perceptions of positive and negative changes resulting from participation in the project. These insights will be important for addressing our proposed research questions related to defining the scope of the proposed interventions, and assessing the feasibility of intervention uptake and implementation. A final project assessment workshop will also be carried out to internally assess the strengths and limitations of the project's M&E framework.

Smoked fish value chains in Ghana have clear potential to influence anemia risk among women fish smokers via multiple, potentially interconnected and contradictory mechanisms. More broadly, these value chains also have significant potential to affect the nutrition and health status of coastal and lake communities and of consumers across the country whose diets are profoundly shaped by these value chains. The investigators expect that the findings of this research will significantly contribute to understanding how best to design, implement, and evaluate interventions into fisheries and other ASF value chains in Ghana and across SSA to address anemia and related nutrition and health concerns.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant
* Not planning to move from the community during the project period
* Engaged in fish processing as primary livelihood

Exclusion Criteria:

* Pregnant
* Planning to move from the community during the project period
* Not engaged in fish processing as primary livelihood

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-08-17 (Actual); Study Completion 2019-08-17 (Actual)

PRIMARY OUTCOMES:
Change in anemia over time | Change from baseline anemia status over the 9 months of the intervention
  Hemoglobin (Hb) <120 g/L, based on analysis of blood and stool samples

SECONDARY OUTCOMES:
Change in knowledge and value of animal-source foods for health over time | Change from baseline knowledge over the 9 months of the intervention
  Evaluated from participants' responses to assessment related to content of audio messages and peer-to-peer learning
Change in amount of processed fish kept for own consumption | Change from baseline amount of fish over the 9 months of the intervention
  Collected daily using participants' business diaries
Change in animal-source food purchases | Change from baseline purchases over the 9 months of the intervention
  Collected using a seven-day animal-source food expenditure questionnaire
Change in consumption of animal-source food | Change from baseline consumption over the 9 months of the intervention
  Collected using a 24-hour dietary recall questionnaire on three non-consecutive days in a one-week period
Change in understanding and valuation of the importance of specific practices for improving environmental and personal hygiene and minimizing risk of infection | Change from baseline understanding over the 9 months of the intervention
  Participant recall and observation of use of insecticide-treated bed nets for sleeping, recent anti-malaria indoor residual spraying of household, frequency and location of barefoot travel, handwashing with soap, safe disposal of stool, treatment of drinking water, safe food and storage preparation practices, and personal hygiene
Change in women's autonomy in decision-making and control over earned income | Change from baseline autonomy over the 9 months of the intervention
  Measure of women's access to productive capital and the role of women in household decision-making related to agricultural production and income generation, as assessed by a questionnaire of the Women's Empowerment in Agriculture Index
Change in smoked fish production and processing capacity | Change from baseline production and capacity over the 9 months of the intervention
  Assessed from daily business diaries and participant recall for cross-validation
Change in fish sales and income generation from fish sales | Change from baseline sales over the 9 months of the intervention
  Assessed from daily business diaries and participant recall for cross-validation
Change in fuelwood and other fish processing business-related expenditures | Change from baseline expenditures over the 9 months of the intervention
  Assessed from daily business diaries and participant recall for cross-validation
Change in knowledge of entrepreneurial skills and best business practices | Change from baseline knowledge and practices over the 9 months of the intervention
  Examined using assessment tool that evaluates knowledge of customer care, calculating profits, managing inventory, and accounting
Change in perceptions of positive and negative changes resulting from participation in interventions | Change from baseline perceptions over the 9 months of the intervention
  Measured from extent to which women used market price information that was disseminated via mobile phones, changes in women's business practices, and women's perceptions of the reasons for changes in fish processing, sales, and/or income from fish sales
Change in exposure to PM2.5 (particulate matter less than 2.5 microns in aerodynamic diameter) and CO (carbon monoxide) | Change from baseline exposure over the 9 months of the intervention
  Primary exposure will be calculated as the mean of recorded concentrations during fish smoking activities (determined by participant time use diaries and corroborated with observational data). Secondary exposure will be calculated as the mean of recorded concentrations during the full 48-hour exposure measurement period
Change in work environments during fish processing including individuals participating in processing activities | Change from baseline environments over the 9 months of the intervention
  Assessed from observation data
Change in knowledge of optimal fish handling and smoking practices for enhancing product quality | Change from baseline knowledge over the 9 months of the intervention
  Assessed using custom tool based on the content of community promotional activities and one-on-one counseling sessions
Change in type of fish smoking oven used | Change from baseline oven used over the 9 months of the intervention
  Assessed from observational data
Women's perceptions of the ease of use of Ahotor oven relative to their prior stoves | At the end of study (10 months)
  Assessed using a semi-structured interview guide through in-person interview with subsample of participants in treatment arm 3
Women's perceptions of the functionality of the new oven | At the end of study (10 months)
  Assessed using a semi-structured interview guide through in-person interview with subsample of participants in treatment arm 3
Differences in home cooking patterns following adoption of new ovens | At the end of study (10 months)
  Assessed using a semi-structured interview guide through in-person interview with subsample of participants in treatment arm 3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana, Legon, Accra, Ghana

REFERENCES:
- [Background] World Health Organization. The global prevalence of anaemia in 2011. Geneva, Switzerland: World Health Organization, 2015.
- [Background] World Health Organization. Worldwide prevalence of anaemia, 1993-2005. Geneva, Switzerland: World Health Organization, 2008.
- [Background] International Food Policy Research Institute. Global Nutrition Report 2016: From Promise to Impact: Ending Malnutrition by 2030. Washington, DC: International Food Policy Research Institute, 2016.
- [Background] Ezzati M, Lopez AD, Rodgers AA, Murray CJL. Comparative quantification of health risks: global and regional burden of disease attributable to selected major risk factors. Geneva, Switzerland: World Health Organization, 2004.
- [Background] Horton S, Ross J. The economics of iron deficiency. Food Policy. 2003;28(1):51-75.
- [Background] Klebanoff MA, Shiono PH, Selby JV, Trachtenberg AI, Graubard BI. Anemia and spontaneous preterm birth. Am J Obstet Gynecol. 1991 Jan;164(1 Pt 1):59-63. doi: 10.1016/0002-9378(91)90626-3. PMID 1986627
- [Background] Scholl TO, Hediger ML, Bendich A, Schall JI, Smith WK, Krueger PM. Use of multivitamin/mineral prenatal supplements: influence on the outcome of pregnancy. Am J Epidemiol. 1997 Jul 15;146(2):134-41. doi: 10.1093/oxfordjournals.aje.a009244. PMID 9230775
- [Background] Zeng L, Dibley MJ, Cheng Y, Dang S, Chang S, Kong L, Yan H. Impact of micronutrient supplementation during pregnancy on birth weight, duration of gestation, and perinatal mortality in rural western China: double blind cluster randomised controlled trial. BMJ. 2008 Nov 7;337:a2001. doi: 10.1136/bmj.a2001. PMID 18996930
- [Background] Christian P, Khatry SK, Katz J, Pradhan EK, LeClerq SC, Shrestha SR, Adhikari RK, Sommer A, West KP Jr. Effects of alternative maternal micronutrient supplements on low birth weight in rural Nepal: double blind randomised community trial. BMJ. 2003 Mar 15;326(7389):571. doi: 10.1136/bmj.326.7389.571. PMID 12637400
- [Background] Rao R, Georgieff MK. Iron in fetal and neonatal nutrition. Semin Fetal Neonatal Med. 2007 Feb;12(1):54-63. doi: 10.1016/j.siny.2006.10.007. Epub 2006 Dec 6. PMID 17157088
- [Background] Stevens GA, Finucane MM, De-Regil LM, Paciorek CJ, Flaxman SR, Branca F, Pena-Rosas JP, Bhutta ZA, Ezzati M; Nutrition Impact Model Study Group (Anaemia). Global, regional, and national trends in haemoglobin concentration and prevalence of total and severe anaemia in children and pregnant and non-pregnant women for 1995-2011: a systematic analysis of population-representative data. Lancet Glob Health. 2013 Jul;1(1):e16-25. doi: 10.1016/S2214-109X(13)70001-9. Epub 2013 Jun 25. PMID 25103581
- [Background] Petry N, Olofin I, Hurrell RF, Boy E, Wirth JP, Moursi M, Donahue Angel M, Rohner F. The Proportion of Anemia Associated with Iron Deficiency in Low, Medium, and High Human Development Index Countries: A Systematic Analysis of National Surveys. Nutrients. 2016 Nov 2;8(11):693. doi: 10.3390/nu8110693. PMID 27827838
- [Background] Balarajan Y, Ramakrishnan U, Ozaltin E, Shankar AH, Subramanian SV. Anaemia in low-income and middle-income countries. Lancet. 2011 Dec 17;378(9809):2123-35. doi: 10.1016/S0140-6736(10)62304-5. Epub 2011 Aug 1. PMID 21813172
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Schumann K, Solomons NW. Perspective: What Makes It So Difficult to Mitigate Worldwide Anemia Prevalence? Adv Nutr. 2017 May 15;8(3):401-408. doi: 10.3945/an.116.013847. Print 2017 May. PMID 28507005
- [Background] Jones AD, Colecraft EK, Awuah RB, Boatemaa S, Lambrecht NJ, Adjorlolo LK, Wilson ML. Livestock ownership is associated with higher odds of anaemia among preschool-aged children, but not women of reproductive age in Ghana. Matern Child Nutr. 2018 Jul;14(3):e12604. doi: 10.1111/mcn.12604. Epub 2018 Apr 2. PMID 29608248
- [Background] Lambrecht NJ, Wilson ML, Jones AD. Assessing the Impact of Animal Husbandry and Capture on Anemia among Women and Children in Low- and Middle-Income Countries: A Systematic Review. Adv Nutr. 2019 Mar 1;10(2):331-344. doi: 10.1093/advances/nmy080. PMID 30854553
- [Background] Nyantakyi-Frompong H, Colecraft E, Awuah R, Boatemaa S, Kushitor M, Adam Y, et al. Leveraging livestock production to address anemia without increasing exposure to adverse health threats: A multisite qualitative study in Ghana. (under review).
- [Background] Pathways to Anemia Prevention Study Team. Pathways to Anemia Prevention Study Field Report. Tamale, Ghana: Innovations for Poverty Action, 2017.
- [Background] Allison EH, Delaporte A, Hellebrandt de Silva D. Integrating fisheries management and aquaculture development with food security and livelihoods for the poor. Report submitted to the Rockefeller Foundation. Norwich, UK: School of International Development, University of East Anglia, 2013.
- [Background] High Level Panel of Experts on Food Security and Nutrition. Sustainable fisheries and aquaculture for food security and nutrition. Rome, Italy: FAO, 2014.
- [Background] Frocklin S, de la Torre-Castro M, Lindstrom L, Jiddawi NS. Fish traders as key actors in fisheries: gender and adaptive management. Ambio. 2013 Dec;42(8):951-62. doi: 10.1007/s13280-013-0451-1. PMID 24213994
- [Background] World Bank. Adwoa Adezawa: The Young Woman and the Sea. Washington, DC: World Bank; 2017 [updated March 22, 2017.
- [Background] Williams SB, editor Economic Potentials of Women in Small-scale Fisheries in West Africa. IIFET 2000 Proceedings; 2000.
- [Background] FAO. The state of world fisheries and aquaculture 2014. Rome, Italy: FAO, 2014.
- [Background] World Bank, FAO, WorldFish. Hidden harvest: the global contribution of capture fisheries. Washington, DC: World Bank, 2012.
- [Background] Koranteng KA. The Ghanaian fishery for sardinellas. In: Bard FX, Koranteng KA, editors. Dynamics and Use of Sardinella Resources from Upwelling off Ghana and Ivory Coast: Acts of DUSRU Meeting. ORSTOM, Colloque DUSRU, 5-8 Oct 1993, Accra, Ghana. Paris, France: ORSTOM Editions; 1995. p. 243-58.
- [Background] Gibson RS, Yeudall F, Drost N, Mtitimuni BM, Cullinan TR. Experiences of a community-based dietary intervention to enhance micronutrient adequacy of diets low in animal source foods and high in phytate: a case study in rural Malawian children. J Nutr. 2003 Nov;133(11 Suppl 2):3992S-3999S. doi: 10.1093/jn/133.11.3992S. PMID 14672301
- [Background] UNDP, FAO. Improved fish smoking: Ghana. In: UNDP, FAO, editors. Sharing Innovative Experiences Volume 5, Examples of Successful Initiatives in Agriculture and Rural Development in the South. Rome, Italy: UNDP, Special Unit for Technical Cooperation among Developing Countries; 2001.
- [Background] Overa R. Partners and Competitors: Gendered Entrepreneurship in Ghanaian Canoe Fisheries: University of Bergen; 1998.
- [Background] Naeher LP, Brauer M, Lipsett M, Zelikoff JT, Simpson CD, Koenig JQ, Smith KR. Woodsmoke health effects: a review. Inhal Toxicol. 2007 Jan;19(1):67-106. doi: 10.1080/08958370600985875. PMID 17127644
- [Background] Fullerton DG, Bruce N, Gordon SB. Indoor air pollution from biomass fuel smoke is a major health concern in the developing world. Trans R Soc Trop Med Hyg. 2008 Sep;102(9):843-51. doi: 10.1016/j.trstmh.2008.05.028. Epub 2008 Jul 17. PMID 18639310
- [Background] Amegah AK, Quansah R, Jaakkola JJ. Household air pollution from solid fuel use and risk of adverse pregnancy outcomes: a systematic review and meta-analysis of the empirical evidence. PLoS One. 2014 Dec 2;9(12):e113920. doi: 10.1371/journal.pone.0113920. eCollection 2014. PMID 25463771
- [Background] Dherani M, Pope D, Mascarenhas M, Smith KR, Weber M, Bruce N. Indoor air pollution from unprocessed solid fuel use and pneumonia risk in children aged under five years: a systematic review and meta-analysis. Bull World Health Organ. 2008 May;86(5):390-398C. doi: 10.2471/blt.07.044529. PMID 18545742
- [Background] Ezzati M, Kammen DM. The health impacts of exposure to indoor air pollution from solid fuels in developing countries: knowledge, gaps, and data needs. Environ Health Perspect. 2002 Nov;110(11):1057-68. doi: 10.1289/ehp.021101057. PMID 12417475
- [Background] Gordon A, Pulis A, Owusu-Adjei E. Smoked marine fish from Western Region, Ghana: a value chain assessment. Ghana: WorldFish Center, USAID Integrated Coastal and Fisheries Governance Initiative for the Western Region, 2011.
- [Background] Béné C, Russell AJM. Diagnostic study of the Volta Basin fisheries, Part 2: Livelihoods and poverty analysis, current trends and projections. Cairo, Egypt: WorldFish Center Regional Offices for Africa and West Asia, 2007.
- [Background] Kamal A, Cincinelli A, Martellini T, Malik RN. A review of PAH exposure from the combustion of biomass fuel and their less surveyed effect on the blood parameters. Environ Sci Pollut Res Int. 2015 Mar;22(6):4076-98. doi: 10.1007/s11356-014-3748-0. Epub 2014 Nov 21. PMID 25410307
- [Background] Prockop LD, Chichkova RI. Carbon monoxide intoxication: an updated review. J Neurol Sci. 2007 Nov 15;262(1-2):122-30. doi: 10.1016/j.jns.2007.06.037. Epub 2007 Aug 27. PMID 17720201
- [Background] Patel A. Household Air Pollution. In: Landrigan PJ, Etzel RA, editors. Textbook of Children's Environmental Health. Oxford, UK: Oxford University Press; 2003.
- [Background] Raub JA, Mathieu-Nolf M, Hampson NB, Thom SR. Carbon monoxide poisoning--a public health perspective. Toxicology. 2000 Apr 7;145(1):1-14. doi: 10.1016/s0300-483x(99)00217-6. PMID 10771127
- [Background] Kelly FJ. Oxidative stress: its role in air pollution and adverse health effects. Occup Environ Med. 2003 Aug;60(8):612-6. doi: 10.1136/oem.60.8.612. No abstract available. PMID 12883027
- [Background] Kampfrath T, Maiseyeu A, Ying Z, Shah Z, Deiuliis JA, Xu X, Kherada N, Brook RD, Reddy KM, Padture NP, Parthasarathy S, Chen LC, Moffatt-Bruce S, Sun Q, Morawietz H, Rajagopalan S. Chronic fine particulate matter exposure induces systemic vascular dysfunction via NADPH oxidase and TLR4 pathways. Circ Res. 2011 Mar 18;108(6):716-26. doi: 10.1161/CIRCRESAHA.110.237560. Epub 2011 Jan 27. PMID 21273555
- [Background] Mishra V, Retherford RD. Does biofuel smoke contribute to anaemia and stunting in early childhood? Int J Epidemiol. 2007 Feb;36(1):117-29. doi: 10.1093/ije/dyl234. Epub 2006 Nov 3. PMID 17085456
- [Background] Sukhsohale ND, Narlawar UW, Phatak MS. Indoor air pollution from biomass combustion and its adverse health effects in central India: an exposure-response study. Indian J Community Med. 2013 Jul;38(3):162-7. doi: 10.4103/0970-0218.116353. PMID 24019602
- [Background] Flintwood-Brace A. Biomass Smoke Exposure in Traditional Smokehouses and Respiratory Symptoms Among Fish Smokers at Aboadze/Abuesi in the Western Region of Ghana: University of Ghana; 2016.
- [Background] Dienye P, Akani A, Okokon I. Respiratory effects of biomass fuel combustion on rural fish smokers in a Nigerian fishing settlement: a case control study. Afr Health Sci. 2016 Jun;16(2):516-23. doi: 10.4314/ahs.v16i2.20. PMID 27605967
- [Background] Ghana Statistical Service, Ghana Health Service, ICF International. Ghana Demographic and Health Survey 2014 Rockville, MD: GSS, GHS, and ICF International, 2015.
- [Background] Beard JL. Iron deficiency: assessment during pregnancy and its importance in pregnant adolescents. Am J Clin Nutr. 1994 Feb;59(2 Suppl):502S-508S discussion 508S-510S. doi: 10.1093/ajcn/59.2.502S. PMID 8304288
- [Background] Barda B, Albonico M, Ianniello D, Ame SM, Keiser J, Speich B, Rinaldi L, Cringoli G, Burioni R, Montresor A, Utzinger J. How long can stool samples be fixed for an accurate diagnosis of soil-transmitted helminth infection using Mini-FLOTAC? PLoS Negl Trop Dis. 2015 Apr 7;9(4):e0003698. doi: 10.1371/journal.pntd.0003698. eCollection 2015 Apr. PMID 25848772
- [Background] Rubin H, Rubin I. Qualitative Interviewing: the Art of Hearing Data. Thousand Oaks, California: Sage; 2005.
- [Background] SPRING, Ghana Health Service. Ghana: Landscape Analysis of Anemia and Anemia Programming. Arlington, VA: Strengthening Partnerships, Results, and Innovations in Nutrition Globally (SPRING) project, 2016.
- [Background] Global Panel on Agriculture and Food Systems for Nutrition. Food systems and diets: Facing the challenges of the 21st century. London, UK: Global Panel on Agriculture and Food Systems for Nutrition, 2016.
- [Background] Haldar K, Mohandas N. Malaria, erythrocytic infection, and anemia. Hematology Am Soc Hematol Educ Program. 2009:87-93. doi: 10.1182/asheducation-2009.1.87. PMID 20008186
- [Background] World Health Organization. Soil-transmitted helminth infections Geneva, Switzerland: World Health Organization; 2017.
- [Background] Yatich NJ, Jolly PE, Funkhouser E, Agbenyega T, Rayner JC, Ehiri JE, Turpin A, Stiles JK, Ellis WO, Jiang Y, Williams JH. The effect of malaria and intestinal helminth coinfection on birth outcomes in Kumasi, Ghana. Am J Trop Med Hyg. 2010 Jan;82(1):28-34. doi: 10.4269/ajtmh.2010.09-0165. PMID 20064991
- [Background] Soares Magalhaes RJ, Biritwum NK, Gyapong JO, Brooker S, Zhang Y, Blair L, Fenwick A, Clements AC. Mapping helminth co-infection and co-intensity: geostatistical prediction in ghana. PLoS Negl Trop Dis. 2011 Jun;5(6):e1200. doi: 10.1371/journal.pntd.0001200. Epub 2011 Jun 7. PMID 21666800
- [Background] Ghana Health Service. National malaria control programme: 2010 Annual Report. Accra, Ghana: Ghana Health Service, 2010.
- [Background] Mockenhaupt FP, Rong B, Gunther M, Beck S, Till H, Kohne E, Thompson WN, Bienzle U. Anaemia in pregnant Ghanaian women: importance of malaria, iron deficiency, and haemoglobinopathies. Trans R Soc Trop Med Hyg. 2000 Sep-Oct;94(5):477-83. doi: 10.1016/s0035-9203(00)90057-9. PMID 11132370
- [Background] Ofori M, Ansah E, Agyepong I, Ofori-Adjei D, Hviid L, Akanmori B. Pregnancy-associated malaria in a rural community of ghana. Ghana Med J. 2009 Mar;43(1):13-8. PMID 19652749
- [Background] Hotez PJ, Bundy DAP, Beegle K, Brooker S, Drake L, de Silva N, Montresor A, Engels D, Jukes M, Chitsulo L, Chow J, Laxminarayan R, Michaud C, Bethony J, Correa-Oliveira R, Shuhua X, Fenwick A, Savioli L. Helminth Infections: Soil-transmitted Helminth Infections and Schistosomiasis. In: Jamison DT, Breman JG, Measham AR, Alleyne G, Claeson M, Evans DB, Jha P, Mills A, Musgrove P, editors. Disease Control Priorities in Developing Countries. 2nd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2006. Chapter 24. Available from http://www.ncbi.nlm.nih.gov/books/NBK11748/ PMID 21250326
- [Background] Naing C, Whittaker MA, Nyunt-Wai V, Reid SA, Wong SF, Mak JW, Tanner M. Malaria and soil-transmitted intestinal helminth co-infection and its effect on anemia: a meta-analysis. Trans R Soc Trop Med Hyg. 2013 Nov;107(11):672-83. doi: 10.1093/trstmh/trt086. PMID 24123127
- [Background] Glanz K, Rimer BK, Viswanath K. Health Behavior and Health Education: Theory, Research, and Practice Edition. San Francisco, CA: Wiley, John & Sons, Inc.; 2008.
- [Background] Manoff Group. Defining Social and Behavior Change Communication and Other Essential Health Communication Terms. Washington, DC: Manoff Group.
- [Background] Sanghvi T, Haque R, Roy S, Afsana K, Seidel R, Islam S, Jimerson A, Baker J. Achieving behaviour change at scale: Alive & Thrive's infant and young child feeding programme in Bangladesh. Matern Child Nutr. 2016 May;12 Suppl 1(Suppl 1):141-54. doi: 10.1111/mcn.12277. PMID 27187912
- [Background] Dewey KG, Adu-Afarwuah S. Systematic review of the efficacy and effectiveness of complementary feeding interventions in developing countries. Matern Child Nutr. 2008 Apr;4 Suppl 1(Suppl 1):24-85. doi: 10.1111/j.1740-8709.2007.00124.x. PMID 18289157
- [Background] Berti PR, Krasevec J, FitzGerald S. A review of the effectiveness of agriculture interventions in improving nutrition outcomes. Public Health Nutr. 2004 Aug;7(5):599-609. doi: 10.1079/PHN2003595. PMID 15251050
- [Background] World Bank. From Agriculture to Nutrition: Pathways, Synergies, and Outcomes Washington, DC: World Bank, 2007.
- [Background] Pathways to Anemia Prevention Study Team. Pathways to Anemia Prevention Study: Report On Results Dissemination and Consensus Building Workshop Accra, Ghana: University of Ghana, 2017.
- [Background] Biran A, Schmidt WP, Varadharajan KS, Rajaraman D, Kumar R, Greenland K, Gopalan B, Aunger R, Curtis V. Effect of a behaviour-change intervention on handwashing with soap in India (SuperAmma): a cluster-randomised trial. Lancet Glob Health. 2014 Mar;2(3):e145-54. doi: 10.1016/S2214-109X(13)70160-8. Epub 2014 Feb 27. PMID 25102847
- [Background] Scott BE, Schmidt WP, Aunger R, Garbrah-Aidoo N, Animashaun R. Marketing hygiene behaviours: the impact of different communication channels on reported handwashing behaviour of women in Ghana. Health Educ Res. 2008 Jun;23(3):392-401. doi: 10.1093/her/cym056. Epub 2007 Nov 13. PMID 18000025
- [Background] Curtis V, Kanki B, Cousens S, Diallo I, Kpozehouen A, Sangare M, Nikiema M. Evidence of behaviour change following a hygiene promotion programme in Burkina Faso. Bull World Health Organ. 2001;79(6):518-27. PMID 11436473
- [Background] Garn JV, Sclar GD, Freeman MC, Penakalapati G, Alexander KT, Brooks P, Rehfuess EA, Boisson S, Medlicott KO, Clasen TF. The impact of sanitation interventions on latrine coverage and latrine use: A systematic review and meta-analysis. Int J Hyg Environ Health. 2017 Apr;220(2 Pt B):329-340. doi: 10.1016/j.ijheh.2016.10.001. Epub 2016 Oct 11. PMID 27825597
- [Background] Freeman MC, Garn JV, Sclar GD, Boisson S, Medlicott K, Alexander KT, Penakalapati G, Anderson D, Mahtani AG, Grimes JET, Rehfuess EA, Clasen TF. The impact of sanitation on infectious disease and nutritional status: A systematic review and meta-analysis. Int J Hyg Environ Health. 2017 Aug;220(6):928-949. doi: 10.1016/j.ijheh.2017.05.007. Epub 2017 May 31. PMID 28602619
- [Background] Ziegelbauer K, Speich B, Mausezahl D, Bos R, Keiser J, Utzinger J. Effect of sanitation on soil-transmitted helminth infection: systematic review and meta-analysis. PLoS Med. 2012 Jan;9(1):e1001162. doi: 10.1371/journal.pmed.1001162. Epub 2012 Jan 24. PMID 22291577
- [Background] Strunz EC, Addiss DG, Stocks ME, Ogden S, Utzinger J, Freeman MC. Water, sanitation, hygiene, and soil-transmitted helminth infection: a systematic review and meta-analysis. PLoS Med. 2014 Mar 25;11(3):e1001620. doi: 10.1371/journal.pmed.1001620. eCollection 2014 Mar. PMID 24667810
- [Background] Waddington H, Snilstveit B, White H, Fewtrell L. Water, sanitation and hygiene interventions to combat childhood diarrhoea in developing countries. Washington, DC: International Initiative for Impact Evaluation (3ie), 2009.
- [Background] Humphrey JH. Child undernutrition, tropical enteropathy, toilets, and handwashing. Lancet. 2009 Sep 19;374(9694):1032-1035. doi: 10.1016/S0140-6736(09)60950-8. No abstract available. PMID 19766883
- [Background] Loll DK, Berthe S, Faye SL, Wone I, Arnold B, Koenker H, Schubert J, Lo Y, Thwing J, Faye O, Weber R. "You need to take care of it like you take care of your soul": perceptions and behaviours related to mosquito net damage, care, and repair in Senegal. Malar J. 2014 Aug 15;13:322. doi: 10.1186/1475-2875-13-322. PMID 25128021
- [Background] Ricotta EE, Boulay M, Ainslie R, Babalola S, Fotheringham M, Koenker H, Lynch M. The use of mediation analysis to assess the effects of a behaviour change communication strategy on bed net ideation and household universal coverage in Tanzania. Malar J. 2015 Jan 21;14:15. doi: 10.1186/s12936-014-0531-0. PMID 25603882
- [Background] Koenker H, Keating J, Alilio M, Acosta A, Lynch M, Nafo-Traore F. Strategic roles for behaviour change communication in a changing malaria landscape. Malar J. 2014 Jan 2;13:1. doi: 10.1186/1475-2875-13-1. PMID 24383426
- [Background] van den Bold M, Quisumbing AR, Gillespie S. Women's Empowerment and Nutrition: An Evidence Review. Washington, DC: International Food Policy Research Institute, 2013.
- [Background] Kennedy E, Cogill B. Income and Nutritional Effects of the Commercialization of Agriculture in Southwestern Kenya. Washington, DC: International Food Policy Research Institute, 1987.
- [Background] Quisumbing AR, Brown L, Feldstein H, Haddad LJ, Pena C. Women: The Key to Food Security. Washington, DC: International Food Policy Research Institute, 1995.
- [Background] The Impact of Non-Traditional Export Agriculture on Income and Food Availability in Guatemala: An Intra-Household Perspective, (1994).
- [Background] Colecraft EK, Marquis GS, Sakyi-Dawson O, Lartey A, Butler LM, Ahunu B, et al. Planning, design and implementation of the enhancing child nutrition through animal source food management (ENAM) project. African Journal of Food, Agriculture, Nutrition and Development. 2012;12(1):5687-708.
- [Background] Sasan A. Mobile Health: A Technology Road Map: Springer; 2015.
- [Background] Farm Radio International. Farmer Radio in Sub-Saharan Africa: A snapshot final report of the African Rural Radio Program Analysis (ARRPA) project. Ottawa, Canada: Farm Radio International, 2014.
- [Background] Ilboudo J-P. After 50 years: The role and use of rural radio in Africa. One to Watch: Radio, New ICTs and Interactivity. Rome, Italy: FAO; 2003.
- [Background] Akapule S. Information Technology Platform Launched in Upper East Region. Ghana News Agency. 2017.
- [Background] SPRING, Ghana Health Service. Health Worker Training Manual for Anaemia Control in Ghana. Accra, Ghana: SPRING and Ghana Health Service, 2017.
- [Background] Lamstein S, Stillman T, Koniz-Booher P, Aakesson A, Collaiezzi B, Williams T, et al. Evidence of Effective Approaches to Social and Behavior Change Communication for Preventing and Reducing Stunting and Anemia: Report from a Systematic Literature Review. Arlington, VA: USAID/Strengthening Partnerships, Results, and Innovations in Nutrition Globally (SPRING) Project, 2014.
- [Background] Aubel J. The roles and influence of grandmothers and men: Evidence supporting a family-focused approach to optimal infant and young child nutrition. Washington, DC: PATH, CARE, Manoff Group, University Research Co., 2011.
- [Background] CARE International. Women's Empowerment and Engaging Men. Atlanta, GA: CARE International, 2009.
- [Background] Gibson RS. Principles of nutritional assessment. New York, NY: Oxford University Press; 2005.
- [Background] International Food Policy Research Institute. Women's empowerment in agriculture index. Washington, DC: International Food Policy Research Institute, 2012.
- [Background] Cho Y, Honorati M. Entrepreneurship Programs in Developing Countries: A Meta Regression Analysis. Washington, DC: World Bank, 2013.
- [Background] International Labor Organization, Women's Entrepreneurship Development Programme. Effectiveness of Entrepreneurship Development Interventions for Women Entrepreneurs. Geneva, Switzerland: International Labor Organization and Women's Entrepreneurship Development Programme, 2015.
- [Background] IFC, G-20 Global Partnership for Financial Inclusion (GPFI). Strengthening access to finance for women-owned small and medium-sized enterprises (SMEs) in developing countries. Washington, DC: GPFI, 2011.
- [Background] De Mel S, McKenzie D, Woodruff C. Business training and female enterprise startup, growth, and dynamics: Experimental evidence from Sri Lanka. Washington, DC: World Bank, 2012.
- [Background] World Bank. World Development Report 2012: Gender Equality and Development. Washington, DC: World Bank, 2011.
- [Background] Hallman K. Mother-Father Resources, Marriage Payments, and Girl-Boy Health in Rural Bangladesh. In: Quisumbing AR, editor. Household Decisions, Gender, and Development. Washington, DC: International Food Policy Research Institute; 2003. p. 115-20.
- [Background] Thomas D. Like Father, Like Son, or Like Mother, Like Daughter: Parental Education and Child Health. Journal of Human Resources. 1994;29(4):950-88.
- [Background] Dima J. Constraints and opportunities facing women entrepreneurs in developing countries: A relational perspective. Gender in Management. 2009;24(4):232-51.
- [Background] Institute for Industrial Research - CSIR, Ghana Standard Authority, Kwarteng E. Testing of Low PAH Improve Fish Smoking Stove (Ahotor oven). Narragansett, RI: USAID/Ghana Sustainable Fisheries Management Project (SFMP), Coastal Resources Center, Graduate School of Oceanography, University of Rhode Island, 2016.
- [Background] Netherlands Development Organization. Introducing the Ahotor oven in the Volta region of Ghana. 2017.
- [Background] Jack DW, Asante KP, Wylie BJ, Chillrud SN, Whyatt RM, Ae-Ngibise KA, Quinn AK, Yawson AK, Boamah EA, Agyei O, Mujtaba M, Kaali S, Kinney P, Owusu-Agyei S. Ghana randomized air pollution and health study (GRAPHS): study protocol for a randomized controlled trial. Trials. 2015 Sep 22;16:420. doi: 10.1186/s13063-015-0930-8. PMID 26395578
- [Background] Quinn AK, Ae-Ngibise KA, Kinney PL, Kaali S, Wylie BJ, Boamah E, Shimbo D, Agyei O, Chillrud SN, Mujtaba M, Schwartz JE, Abdalla M, Owusu-Agyei S, Jack DW, Asante KP. Ambulatory monitoring demonstrates an acute association between cookstove-related carbon monoxide and blood pressure in a Ghanaian cohort. Environ Health. 2017 Jul 21;16(1):76. doi: 10.1186/s12940-017-0282-9. PMID 28732501
- [Background] Rodes CE, Chillrud SN, Haskell WL, Intille SS, Albinali F, Rosenberger M. Predicting Adult Pulmonary Ventilation Volume and Wearing Compliance by On-Board Accelerometry During Personal Level Exposure Assessments. Atmos Environ (1994). 2012 Sep;57:126-137. doi: 10.1016/j.atmosenv.2012.03.057. PMID 24065872
- [Background] Quansah R, Semple S, Ochieng CA, Juvekar S, Armah FA, Luginaah I, Emina J. Effectiveness of interventions to reduce household air pollution and/or improve health in homes using solid fuel in low-and-middle income countries: A systematic review and meta-analysis. Environ Int. 2017 Jun;103:73-90. doi: 10.1016/j.envint.2017.03.010. Epub 2017 Mar 22. PMID 28341576
- [Background] World Health Organization. Haemoglobin concentrations for the diagnosis of anaemia and assessment of severity. Geneva, Switzerland: World Health Organization, 2011.
- [Background] Erhardt JG, Estes JE, Pfeiffer CM, Biesalski HK, Craft NE. Combined measurement of ferritin, soluble transferrin receptor, retinol binding protein, and C-reactive protein by an inexpensive, sensitive, and simple sandwich enzyme-linked immunosorbent assay technique. J Nutr. 2004 Nov;134(11):3127-32. doi: 10.1093/jn/134.11.3127. PMID 15514286
- [Background] Yap P, Furst T, Muller I, Kriemler S, Utzinger J, Steinmann P. Determining soil-transmitted helminth infection status and physical fitness of school-aged children. J Vis Exp. 2012 Aug 22;(66):e3966. doi: 10.3791/3966. PMID 22951972
- [Background] Namaste SM, Rohner F, Huang J, Bhushan NL, Flores-Ayala R, Kupka R, Mei Z, Rawat R, Williams AM, Raiten DJ, Northrop-Clewes CA, Suchdev PS. Adjusting ferritin concentrations for inflammation: Biomarkers Reflecting Inflammation and Nutritional Determinants of Anemia (BRINDA) project. Am J Clin Nutr. 2017 Jul;106(Suppl 1):359S-371S. doi: 10.3945/ajcn.116.141762. Epub 2017 Jun 14. PMID 28615259
- [Background] Larson LM, Addo OY, Sandalinas F, Faigao K, Kupka R, Flores-Ayala R, Suchdev PS. Accounting for the influence of inflammation on retinol-binding protein in a population survey of Liberian preschool-age children. Matern Child Nutr. 2017 Apr;13(2):e12298. doi: 10.1111/mcn.12298. Epub 2016 Feb 4. PMID 26842430
- [Background] Corbin J, Strauss A. Grounded theory research: procedures, canons, and evaluative criteria. Qualitative Sociology. 1990;13(1):3e21.
- [Background] Stoltzfus RJ. Iron interventions for women and children in low-income countries. J Nutr. 2011 Apr 1;141(4):756S-762S. doi: 10.3945/jn.110.128793. Epub 2011 Mar 2. PMID 21367936
- [Background] World Health Organization. Iron supplementation during pregnancy: why aren't women complying? Geneva, Switzerland: World Health Organization, 1990.
- [Background] Schultink W, van der Ree M, Matulessi P, Gross R. Low compliance with an iron-supplementation program: a study among pregnant women in Jakarta, Indonesia. Am J Clin Nutr. 1993 Feb;57(2):135-9. doi: 10.1093/ajcn/57.2.135. PMID 8424380
- [Background] Girard AW, Self JL, McAuliffe C, Olude O. The effects of household food production strategies on the health and nutrition outcomes of women and young children: a systematic review. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:205-22. doi: 10.1111/j.1365-3016.2012.01282.x. PMID 22742612
- [Background] Leroy JL, Frongillo EA. Can interventions to promote animal production ameliorate undernutrition? J Nutr. 2007 Oct;137(10):2311-6. doi: 10.1093/jn/137.10.2311. PMID 17885016
- [Background] Hall SJ, Hilborn R, Andrew NL, Allison EH. Innovations in capture fisheries are an imperative for nutrition security in the developing world. Proc Natl Acad Sci U S A. 2013 May 21;110(21):8393-8. doi: 10.1073/pnas.1208067110. Epub 2013 May 13. PMID 23671089
- [Background] Kawarazuka N, Bene C. The potential role of small fish species in improving micronutrient deficiencies in developing countries: building evidence. Public Health Nutr. 2011 Nov;14(11):1927-38. doi: 10.1017/S1368980011000814. Epub 2011 May 20. PMID 21729489
- [Background] Herforth A, Jones A, Pinstrup-Andersen P. Prioritizing Nutrition in Agriculture and Rural Development: Guiding Principles for Operational Investments. Washington, DC: World Bank, 2012.
- [Background] Jones AD. Healthy Food for a Healthy World: Leveraging Agriculture and Food to Improve Global Nutrition. Chicago, IL: Chicago Council on Global Affairs, 2015.
- [Background] Marquis GS, Colecraft EK. The Nutrition-Microcredit Synergy: A Case For Multiple Interventions and Strategies. African Journal of Food, Agriculture, Nutrition and Development. 2012;12(1):5674-86.
- [Background] Homiah PA, Sakyi-Dawson O, Bonsu AM, Marquis GS. Microenterprise development coupled with nutrition education can help increase caregivers' incomes and household accessibility to animal source foods. African Journal of Food, Agriculture, Nutrition and Development. 2012;12(1):5725-45.
- [Background] Santarelli RL, Pierre F, Corpet DE. Processed meat and colorectal cancer: a review of epidemiologic and experimental evidence. Nutr Cancer. 2008;60(2):131-44. doi: 10.1080/01635580701684872. PMID 18444144
- [Background] Farrow DC, Vaughan TL, Berwick M, Lynch CF, Swanson GM, Lyon JL. Diet and nasopharyngeal cancer in a low-risk population. Int J Cancer. 1998 Dec 9;78(6):675-9. doi: 10.1002/(sici)1097-0215(19981209)78:63.0.co;2-j. PMID 9833758
- See also: International Food Policy Research Institute. Women's Empowerment in Agriculture Index. — http://www.ifpri.org/publication/womens-empowerment-agriculture-index
- See also: Netherlands Development Organization. Introducing the Ahotor oven in the Volta region of Ghana. 2017. — http://www.snv.org/update/introducing-ahotor-oven-volta-region-ghana